CLINICAL TRIAL: NCT04462861
Title: A New Securement Method for External Tunneled Central Venous Access Devices (CVAD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-1592
Record Dates: First submitted 2020-06-24; First posted 2020-07-08 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Central Venous Catheter Exit Site Infection; Central Venous Catheter Related Bloodstream Infection
Keywords: central venous access device, CVAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CVAD securement device (Experimental): Patients with a pre-existing CVAD who will trial the new securement dressing
  Interventions: Device: Central venous access device (CVAD) Snuggie Securement Device

INTERVENTIONS:
Device: Central venous access device (CVAD) Snuggie Securement Device — Participants will be given a prototype of a CVAD securement device for a three week trial. Descriptive data relating to user satisfaction will be collected at 1 and 3 weeks

SUMMARY:
An external tunneled central venous access device (CVAD) is a small plastic tube that is tunneled under the skin into a major vein for long-term use (Figure 1). Patients who require a tunneled CVAD are some of the sickest patients we encounter and include oncology, hematology, and gastrointestinal (intestinal failure) patients. These patients are heavily reliant on their tunneled CVAD, which can be a lifeline for long-term administration of chemotherapeutics, IV medications, blood product transfusions, antibiotics, enteral nutrition, blood draws and fluids. Unfortunately, nearly 30% of pediatric external tunneled CVADs fail prior to the completion of treatment. External tunneled CVAD failures lead to unnecessary morbidity and mortality, interruption of medical therapy, and the added costs and risks associated with additional procedural complications. It is hypothesized that a newly designed securement method for external tunneled central venous access devices (CVAD) will reduce catheter-related complications and increase patient, parent and provider satisfaction, compared to the current standard of care, which is a clear transparent film dressing over the catheter exit site. A 20 patient, prospective clinical trial is proposed to address the following specific aims, which will determine if the securement device:

1. Is rated by patients, parents and providers as easy to apply and comfortable for users
2. Reduces CVAD-related complications, such as delayed healing of the tract, catheter-related infections, and episodes of catheter dislodgement
3. Improves the quality of life for patients and their parents
4. Is preferred over the standard, clear transparent dressing alone
5. Requires any design modifications to improve performance and/or comfort of the device

DETAILED DESCRIPTION:
A prospective pilot trial to examine the feasibility for a new CVAD securement device prototype (see appendix for computer-aided design drawings). Eligible patients will be identified by either mid-level providers, consulting services, or attending surgeons. Researchers will obtain consent from the patient or their parent/legal guardian. Caregivers will be educated on how to apply the securement device and will be given a number to call should they have any questions or concerns. Once the patient is enrolled and provided with the device, the investigators will perform follow up telephone interviews at one and three weeks to evaluate their experience and ensure they did not experience any adverse events.

The investigators will prospectively record the primary and secondary outcomes regarding use of the securement device, including: comfort, quality of materials, adhesive, ease of use, skin problems, infections, dislodgement episodes, catheter breakage, types and numbers of interactions with healthcare providers (phone calls, emergency department and clinic visits), perceived safety, and overall impressions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 31 days to 18 years old, who will undergo surgical placement of a tunneled CVAD
* Any patient with a pre-existing CVAD, who presents to the surgery clinic, emergency department, or is seen as an inpatient consult relating to complications associated with their CVAD
* Patients admitted to the hospital with a pre-existing CVAD for reasons unrelated to the CVAD will be eligible for the study

Exclusion Criteria:

* Any assenting child or consenting parent/guardian can at any time refuse to participate in the study and will be removed
* Any patient whose parents or legal guardians cannot be reached in person or by telephone to provide consent
* Any prisoners, pregnant women, or person with impaired decision-making capacity

Ages: 31 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Comfort | 3 weeks
  Survey question asking for qualitative description of satisfaction
quality of materials | 3 weeks
  Survey question asking for qualitative description of satisfaction
Quality of Adhesive | 3 weeks
  Survey question asking for qualitative description of satisfaction
Ease of use | 3 weeks
  Survey question asking for qualitative description of satisfaction
Skin irritation | 3 weeks
  Survey question asking for qualitative description of complication, if applicable
Infection | 3 weeks
  Survey question asking for qualitative description of complication, if applicable
dislodgement | 3 weeks
  Survey question asking for qualitative description of complication, if applicable
catheter breakage | 3 weeks
  Survey question asking for qualitative description of complication, if applicable
types and numbers of interactions with healthcare providers | 3 weeks
  Survey question asking for qualitative description of interaction, if applicable
Perceived safety | 3 weeks
  Survey question asking for qualitative description of perceived device safety
overall impression | 3 weeks
  Survey question asking for qualitative description of overall impression of device

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Moulton, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Background] Ullman AJ, Marsh N, Mihala G, Cooke M, Rickard CM. Complications of Central Venous Access Devices: A Systematic Review. Pediatrics. 2015 Nov;136(5):e1331-44. doi: 10.1542/peds.2015-1507. Epub 2015 Oct 12. PMID 26459655
- [Background] Ullman AJ, Cooke M, Rickard C. Examining the role of securement and dressing products to prevent central venous access device failure: a narrative review J Assoc Vasc Access 2015; 20:99-110
- [Background] Frey AM, Schears GJ. Why are we stuck on tape and suture? A review of catheter securement devices. J Infus Nurs. 2006 Jan-Feb;29(1):34-8. doi: 10.1097/00129804-200601000-00007. PMID 16428999
- [Background] Orgel E, Ji L, Pastor W, Schore RJ. Infectious morbidity by catheter type in neutropenic children with cancer. Pediatr Infect Dis J. 2014 Mar;33(3):263-6. doi: 10.1097/INF.0000000000000060. PMID 24263218
- [Background] Brandt B, DePalma J, Irwin M, Shogan J, Lucke JF. Comparison of central venous catheter dressings in bone marrow transplant recipients. Oncol Nurs Forum. 1996 Jun;23(5):829-36. PMID 8792352
- [Background] Shivnan JC, McGuire D, Freedman S, Sharkazy E, Bosserman G, Larson E, Grouleff P. A comparison of transparent adherent and dry sterile gauze dressings for long-term central catheters in patients undergoing bone marrow transplant. Oncol Nurs Forum. 1991 Nov-Dec;18(8):1349-56. PMID 1762975
- [Background] Chambers ST, Sanders J, Patton WN, Ganly P, Birch M, Crump JA, Spearing RL. Reduction of exit-site infections of tunnelled intravascular catheters among neutropenic patients by sustained-release chlorhexidine dressings: results from a prospective randomized controlled trial. J Hosp Infect. 2005 Sep;61(1):53-61. doi: 10.1016/j.jhin.2005.01.023. PMID 16002181
- [Background] Ruschulte H, Franke M, Gastmeier P, Zenz S, Mahr KH, Buchholz S, Hertenstein B, Hecker H, Piepenbrock S. Prevention of central venous catheter related infections with chlorhexidine gluconate impregnated wound dressings: a randomized controlled trial. Ann Hematol. 2009 Mar;88(3):267-72. doi: 10.1007/s00277-008-0568-7. Epub 2008 Aug 5. PMID 18679683
- [Background] Ullman AJ, Kleidon T, Gibson V, McBride CA, Mihala G, Cooke M, Rickard CM. Innovative dressing and securement of tunneled central venous access devices in pediatrics: a pilot randomized controlled trial. BMC Cancer. 2017 Aug 30;17(1):595. doi: 10.1186/s12885-017-3606-9. PMID 28854967